CLINICAL TRIAL: NCT03060044
Title: Pharmacokinetic Study Comparing Salmeterol/Fluticasone Easyhaler Products and Seretide Diskus 50/500 µg/Inhalation: A Randomised, Open, Single Centre, Single Dose, Crossover Study in Healthy Subjects
Brief Title: Pharmacokinetic Study Comparing Salmeterol/Fluticasone Easyhaler and Seretide Diskus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3106010
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2016-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Salmeterol Xinafoate; Charcoal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Salmeterol/fluticasone Easyhaler (Experimental): single dose of Salmeterol/fluticasone Easyhaler
  Interventions: Drug: Salmeterol/fluticasone Easyhaler
- Salmeterol/fluticasone Easyhaler with charcoal (Experimental): Single dose of Salmeterol/fluticasone Easyhaler with concomitant charcoal administration
  Interventions: Drug: Salmeterol/fluticasone Easyhaler with charcoal
- Seretide Diskus (Active Comparator): Single dose of Seretide Diskus
  Interventions: Drug: Seretide Diskus
- Seretide Diskus with charcoal (Active Comparator): Single dose of Seretide Diskus with concomitant charcoal administration
  Interventions: Drug: Seretide Diskus with charcoal

INTERVENTIONS:
Drug: Salmeterol/fluticasone Easyhaler
  Arms: Salmeterol/fluticasone Easyhaler
Drug: Salmeterol/fluticasone Easyhaler with charcoal
  Arms: Salmeterol/fluticasone Easyhaler with charcoal
Drug: Seretide Diskus
  Arms: Seretide Diskus
Drug: Seretide Diskus with charcoal
  Arms: Seretide Diskus with charcoal

SUMMARY:
Pharmacokinetic study comparing Salmeterol/fluticasone Easyhaler products and Seretide Diskus 50/500 µg/inhalation; a randomised, open, single centre, single dose, crossover study in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* written informed consent obtained
* good general health ascertained by detailed medical history, and laboratory and physical examinations

Exclusion Criteria:

* evidence of a clinically significant cardiovascular, renal, hepatic, hematological, GI, pulmonary, metabolic-endocrine, neurological or psychiatric disease within the previous 2 years
* any condition requiring concomitant treatment (including vitamins and herbal products)or likely to need any concomitant treatment during the study. as an exception paracetamol and ibuprofen for occasional pain are allowed
* known hypersensitivity to the active substance(s) or the excipient (lactose, which contains small amounts of milk protein) of the drug
* pregnant or lactating females

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Cmax of plasma salmeterol and fluticasone propionate | 0 hour to 34 hours after study treatment administration
AUCt of plasma salmeterol and fluticasone propionate | 0 hour to 34 hours after study treatment administration

CONTACTS AND LOCATIONS:
Overall Officials: Iissa Kivistö, Study Director — Clinical Study director
Locations (1):
- Orion Pharma pharmacology Unit, Espoo, Finland

IPD SHARING:
Plan to Share IPD: Undecided